CLINICAL TRIAL: NCT01823718
Title: Cell Bank of Epstein Barr Virus Specific Cytotoxic T Lymphocytes
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04/7-M
Record Dates: First submitted 2013-03-29; First posted 2013-04-04 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-03

CONDITIONS: EBV Associated Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Injection of allogenic CTL EBV specific

SUMMARY:
Patients patients enrolled in this study have a Lymphoma caused by EBV (after bone marrow transplantation, organ transplantation or patient immunodeficient.

They will receive one to three injections of allogenic CTL specific EBV.

The purpose of this study is to ensure that these injections can not cause a GVH and to study what the side effects are and to see whether this therapy might help patients with Lymphoma.

Immunological monitoring will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, without immunosuppressed organ transplant or immunocompromised and who received a kidney transplant, or kidney-pancreas, or heart or lung or heart-lung, or liver, or cells hematopoietic stem cells, and has given its consent
* Aged 18 to 75 years Children aged more than 12 months,
* PS <4
* Viral load determined EBV
* Life expectancy> 1 month
* Patient typed for HLA DP DQ DR ABC
* Patients with lymphoma in the immunosuppressed associated with EBV and failure, partial response (<50%) or relapsed after treatment with monoclonal antibodies and / or chemotherapy completed for at least three weeks. Patients with partial response may have a PET scan to confirm the lack of response.
* Patient with a measurable mass to assess the response or bone marrow infiltration and / or measurable blood and having frozen tumor material or having a repeat biopsy.
* Availability of a CTL matching at least two HLA or one HLA after validation experts with tumor cells
* test de cytotoxicity negative

Exclusion Criteria:

* Patient Pregnant or lactating
* Concurrent infection with HIV
* EBV negative lymphomas
* If acute GVHD> grade II J-1 before injection (case grafts CSH)
* Treatment of molecules in pre-marketing authorization older than 21 days
* No matching at least two CTL HLA or non expert validation for the use of CTL with HLA sharing a single tumor
* Test of cytotoxicity positive
* Lack of recognition of tumor cells when available

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2007-02; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
The safety of one to three injections of allogenic EBV specific CTLs will be determined through adverse event measurement | 3 months post last injection

SECONDARY OUTCOMES:
To determine the survival, and anti-tumor effects of EBV specific cytotoxic T-lymphocyte lines. | 1 year

OTHER OUTCOMES:
biological monitoring | 12 months

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - CHU de Bordeaux, Bordeaux
  - CHU de Brest, Brest
  - CHU de Lille, Lille
  - CHU de Limoges, Limoges
  - CHU de Nantes, Nantes
  - Hopital Pitié Salpétrière, Paris
  - Hôpital Necker, Paris

REFERENCES:
- [Derived] Gallot G, Vollant S, Saiagh S, Clemenceau B, Vivien R, Cerato E, Bignon JD, Ferrand C, Jaccard A, Vigouroux S, Choquet S, Dalle JH, Frachon I, Bruno B, Mothy M, Mechinaud F, Leblond V, Milpied N, Vie H. T-cell therapy using a bank of EBV-specific cytotoxic T cells: lessons from a phase I/II feasibility and safety study. J Immunother. 2014 Apr;37(3):170-9. doi: 10.1097/CJI.0000000000000031. PMID 24598452